CLINICAL TRIAL: NCT04756531
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO CONTROLLED, SINGLE- AND MULTIPLE-DOSE ESCALATION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF PF 07321332 IN HEALTHY ADULT PARTICIPANTS
Brief Title: STUDY OF PF-07321332 IN HEALTHY PARTICIPANTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: C4671001; 2020-006073-30 (EudraCT Number)
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- PF-07321332 Dose 1 (Experimental): Dose level 1 of PF-07321332
  Interventions: Drug: PF-07321332 Dose 1
- PF-07321332 Dose 2 (Experimental): Dose level 2 of PF-07321332
  Interventions: Drug: PF-07321332 Dose 2
- PF-07321332 Dose 3 (Experimental): Dose level 3 of PF-07321332
  Interventions: Drug: PF-07321332 Dose 3
- PF-07321332 Dose 4 (Experimental): Dose level 4 of PF-07321332
  Interventions: Drug: PF-07321332 Dose 4
- PF-07321332 Dose 5 (Experimental): Dose level 5 of PF-07321332
  Interventions: Drug: PF-07321332 Dose 5
- PF-07321332 Dose 4 (Fed) (Experimental): Dose level 4 of PF-07321332 with high fat meal
  Interventions: Drug: PF-07321332 Dose 4 or Placebo (Fed)

INTERVENTIONS:
Drug: PF-07321332 Dose 1 — PF-07321332 Dose 1 or Placebo
  Arms: PF-07321332 Dose 1
Drug: PF-07321332 Dose 2 — PF-07321332 Dose 2 or Placebo
  Arms: PF-07321332 Dose 2
Drug: PF-07321332 Dose 3 — PF-07321332 Dose 3 or Placebo
  Arms: PF-07321332 Dose 3
Drug: PF-07321332 Dose 4 — PF-07321332 Dose 4 or Placebo
  Arms: PF-07321332 Dose 4
Drug: PF-07321332 Dose 5 — PF-07321332 Dose 5 or Placebo
  Arms: PF-07321332 Dose 5
Drug: PF-07321332 Dose 4 or Placebo (Fed) — PF-07321332 Dose 5 or Placebo with high fat meal
  Arms: PF-07321332 Dose 4 (Fed)

SUMMARY:
A Phase 1, double blind, sponsor open, single and multiple ascending dose study to evaluate safety, tolerability and pharmacokinetics of PF-07321332 in healthy participants.

DETAILED DESCRIPTION:
Combined 5-part study. Part-1: Single Ascending dose Part-2: Multiple Ascending Dose Part-3: Relative bioavailability and food effect Part-4: Metabolism and Excretion Part-5: Supra-therapeutic Exposure Part-1,2 and 5 are double blind, sponsor open and Part-3 and 4 are open label study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between ages of 18-60 years. Male only in part-4.
* Body Mass Index (BMI) of 17.5 to 30.5kg/m2; and a total body weight >50kg (110lbs)
* Japanese subjects who have four Japanese biologic grandparents born in Japan

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy, intestinal resection).
* Positive test result for SARS-CoV-2 infection at the time of screening or Day-1.
* Have received COVID-19 vaccine within 7 days before screening or have received only one of the 2 required doses of COVID-19 vaccine
* Use of tobacco or nicotine containing products in excess of the equivalents of 5 cigarettes per day or 2 chews of tobacco per day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Singh RSP, Toussi SS, Hackman F, Chan PL, Rao R, Allen R, Van Eyck L, Pawlak S, Kadar EP, Clark F, Shi H, Anderson AS, Binks M, Menon S, Nucci G, Bergman A. Innovative Randomized Phase I Study and Dosing Regimen Selection to Accelerate and Inform Pivotal COVID-19 Trial of Nirmatrelvir. Clin Pharmacol Ther. 2022 Jul;112(1):101-111. doi: 10.1002/cpt.2603. Epub 2022 May 4. PMID 35388471
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 5-part study combining PART-1: single ascending dose (SAD), PART-2: multiple ascending dose (MAD), PART-3: relative bioavailability/food effect (rBA/FE), PART-4: metabolism and excretion (M&E) and PART-5: supratherapeutic exposure (SE).
Groups:
- PART-1: SAD Treatment Sequence 1: PF-07321332 150 mg (Suspension), Fasted=>PF-07321332 1500 mg (Suspension), Fasted=>Placebo (Suspension)/ritonavir (RTV) 100 mg, Fasted Participants received a single dose of PF-07321332 150 mg under fasted condition in period 1, a single dose of PF-07321332 1500 mg under fasted condition in period 2, a single dose of placebo and a total of 3 doses of RTV 100 mg at -12h, 0h and 12h post-dose under fasted condition in period 3. There was a washout interval of ≥5 days between periods.
- PART-1: SAD Treatment Sequence 2: PF-07321332 150 mg (Suspension), Fasted=>Placebo (Suspension), Fasted=>PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted Participants received a single dose of PF-07321332 150 mg under fasted condition in period 1, a single dose of placebo under fasted condition in period 2, a single dose of PF-07321332 750 mg and a total of 3 doses of RTV 100 mg at -12h, 0h and 12h post-dose under fasted condition in period 3. There was a washout interval of ≥5 days between periods.
- PART-1:SAD Treatment Sequence 3: Placebo (Suspension), Fasted=>PF-07321332 1500 mg (Suspension), Fasted=>PF-07321332 750 mg (suspension)/RTV 100 mg, Fasted Participants received a single dose of placebo under fasted condition in period 1, a single dose of PF-07321332 1500 mg under fasted condition in period 2, a single dose of PF-07321332 750 mg and a total of 3 doses of RTV 100 mg at -12 hour (h), 0h and 12h post-dose under fasted condition in period 3. There was a washout interval of ≥5 days between periods.
- PART-1: SAD Treatment Sequence 4: PF-07321332 500 mg (Suspension), Fasted=>PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted=>PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed Participants received a single dose of PF-07321332 500 mg under fasted condition in period 1, a single dose of PF-07321332 250 mg and a total of 3 doses of RTV 100 mg at -12h, 0h and 12h post-dose under fasted condition in period 2, a single dose of PF-07321332 250 mg and a total of 3 doses of RTV 100 mg at -12h, 0h and 12h post-dose under fed condition in period 3. There was a washout interval of ≥5 days between periods.
- PART-1: SAD Treatment Sequence 5: PF-07321332 500 mg (Suspension), Fasted=>Placebo (Suspension)/RTV 100 mg, Fasted=>Placebo (Suspension)/RTV 100 mg, Fed Participants received a single dose of PF-07321332 500 mg under fasted condition in period 1, a single dose of placebo and a total of 3 doses of RTV 100 mg at -12h, 0h and 12h post-dose under fasted condition in period 2, a single dose of placebo and a total of 3 doses of RTV 100 mg at -12h, 0h and 12h post-dose under fed condition in period 3. There was a washout interval of ≥5 days between periods.
- PART-1: SAD Treatment Sequence 6: Placebo (Suspension), Fasted=>PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted=>PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed Participants received a single dose of placebo under fasted condition in period 1, a single dose of PF-07321332 250 mg and a total of 3 doses of RTV 100 mg at -12h, 0h and 12h post-dose under fasted condition in period 2, a single dose of PF-07321332 250 mg and a total of 3 doses of RTV 100 mg at -12h, 0h and 12h post-dose under fed condition in period 3. There was a washout interval of ≥5 days between periods.
- PART-2: MAD Placebo (Suspension)/RTV 100 mg Twice Daily (BID), Fasted: Participants received placebo and RTV 100 mg BID under fasted condition for 10 days.
- PART-2: MAD PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted: Participants received PF-07321332 75 mg and RTV 100 mg BID under fasted condition for 10 days.
- PART-2: MAD PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted: Participants received PF-07321332 250 mg and RTV 100 mg BID under fasted condition for 10 days.
- PART-2: MAD PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted: Participants received PF-07321332 500 mg and RTV 100 mg BID under fasted condition for 10 days.
- PART-2: MAD Placebo (Suspension)/RTV100 mg BID, Fasted, Japanese: Japanese participants received placebo and RTV 100 mg BID under fasted condition for 10 days.
- PART-2: MAD PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese: Japanese participants received PF-07321332 250 mg and RTV 100 mg BID under fasted condition for 10 days.
- PART-3: rBA/FE Treatment Sequence 1: PF-07321332 250 mg (Suspension), Fasted=>PF-07321332 250 mg (Tablet), Fasted=>PF-07321332 250 mg (Tablet), Fed Participants received a single dose of PF-07321332 250 mg (suspension) under fasted condition in period 1, PF-07321332 250 mg (tablet) under fasted condition in period 2, and PF-07321332 250 mg (tablet) under fed condition in period 3. There was a washout interval of at least 2 days between dosing in each period.
- PART-3: rBA/FE Treatment Sequence 2: PF-07321332 250 mg (Tablet), Fasted=>PF-07321332 250 mg (Tablet), Fed=>PF-07321332 250 mg (Suspension), Fasted Participants received a single dose of PF-07321332 250 mg (tablet) under fasted condition in period 1, PF-07321332 250 mg (tablet) under fed condition in period 2, and PF-07321332 250 mg (suspension) under fasted condition in period 3. There was a washout interval of at least 2 days between dosing in each period.
- PART-3: rBA/FE Treatment Sequence 3: PF-07321332 250 mg (Tablet), Fed=>PF-07321332 250 mg (Suspension), Fasted=>PF-07321332 250 mg (Tablet), Fasted Participants received a single dose of PF-07321332 250 mg (tablet) under fed condition in period 1, PF-07321332 250 mg (suspension) under fasted condition in period 2, and PF-07321332 250 mg (tablet) under fasted condition in period 3. There was a washout interval of at least 2 days between dosing in each period.
- PART-4: M&E PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted: Participants received a single oral dose of PF-07321332 300 mg with RTV (4 doses of 100 mg at -12h, 0h, 12h, and 24h relative to PF-07321332) under fasted condition.
- PART-5: SE Placebo (Suspension)/RTV 100 mg=>PF-07321332 2250 mg (Suspension)/RTV 100 mg: In period 1, participants received placebo (3 split doses at 0, 2h, and 4h) with RTV (3 doses of 100 mg at -12h, 0h and 12h post-dose) approximately 2h after breakfast. In period 2, participants received PF-07321332 2250 mg (divided into 3 doses of 750 mg administered at 0, 2h, and 4h) with RTV (3 doses of 100 mg at -12h, 0h and 12h post-dose) approximately 2h after breakfast. There was a washout interval of ≥5 days between periods.
- PART-5: SE PF-07321332 2250 mg (Suspension)/RTV 100 mg=>Placebo (Suspension)/RTV 100 mg: In period 1, participants received PF-07321332 2250 mg (divided into 3 doses of 750 mg administered at 0, 2h, and 4h) with RTV (3 doses of 100 mg at -12h, 0h and 12h post-dose) approximately 2h after breakfast. In period 2, participants received placebo (3 split doses at 0, 2h, and 4h) with RTV (3 doses of 100 mg at -12h, 0h and 12h post-dose) approximately 2h after breakfast. There was a washout interval of ≥5 days between periods.
Period: Overall Study
Arm/Group | PART-1: SAD Treatment Sequence 1 | PART-1: SAD Treatment Sequence 2 | PART-1:SAD Treatment Sequence 3 | PART-1: SAD Treatment Sequence 4 | PART-1: SAD Treatment Sequence 5 | PART-1: SAD Treatment Sequence 6 | PART-2: MAD Placebo (Suspension)/RTV 100 mg Twice Daily (BID), Fasted | PART-2: MAD PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PART-2: MAD PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PART-2: MAD PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PART-2: MAD Placebo (Suspension)/RTV100 mg BID, Fasted, Japanese | PART-2: MAD PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese | PART-3: rBA/FE Treatment Sequence 1 | PART-3: rBA/FE Treatment Sequence 2 | PART-3: rBA/FE Treatment Sequence 3 | PART-4: M&E PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted | PART-5: SE Placebo (Suspension)/RTV 100 mg=>PF-07321332 2250 mg (Suspension)/RTV 100 mg | PART-5: SE PF-07321332 2250 mg (Suspension)/RTV 100 mg=>Placebo (Suspension)/RTV 100 mg
Started | 2 | 2 | 2 | 2 | 3 | 2 | 8 | 4 | 4 | 7 | 2 | 4 | 4 | 4 | 4 | 6 | 5 | 5
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 4 | 4 | 7 | 2 | 4 | 4 | 4 | 4 | 6 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled in the study.
Groups:
- PART-1: SAD Treatment Sequence 1: PF-07321332 150 mg (Suspension), Fasted=>PF-07321332 1500 mg (Suspension), Fasted=>Placebo (Suspension)/RTV 100 mg, Fasted Participants received a single dose of PF-07321332 150 mg under fasted condition in period 1, a single dose of PF-07321332 1500 mg under fasted condition in period 2, a single dose of placebo and a total of 3 doses of RTV 100 mg at -12h, 0h and 12h post-dose under fasted condition in period 3. There was a washout interval of ≥5 days between periods.
- Total: Total of all reporting groups
Arm/Group | PART-1: SAD Treatment Sequence 1 | PART-1: SAD Treatment Sequence 2 | PART-1:SAD Treatment Sequence 3 | PART-1: SAD Treatment Sequence 4 | PART-1: SAD Treatment Sequence 5 | PART-1: SAD Treatment Sequence 6 | PART-2: MAD Placebo (Suspension)/RTV 100 mg Twice Daily (BID), Fasted | PART-2: MAD PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PART-2: MAD PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PART-2: MAD PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PART-2: MAD Placebo (Suspension)/RTV100 mg BID, Fasted, Japanese | PART-2: MAD PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese | PART-3: rBA/FE Treatment Sequence 1 | PART-3: rBA/FE Treatment Sequence 2 | PART-3: rBA/FE Treatment Sequence 3 | PART-4: M&E PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted | PART-5: SE Placebo (Suspension)/RTV 100 mg=>PF-07321332 2250 mg (Suspension)/RTV 100 mg | PART-5: SE PF-07321332 2250 mg (Suspension)/RTV 100 mg=>Placebo (Suspension)/RTV 100 mg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 2 | 8 | 4 | 4 | 7 | 2 | 4 | 4 | 4 | 4 | 6 | 5 | 5 | 70
Age, Customized [Number; unit: Participants]
  18-44 Years | 0 | 1 | 2 | 2 | 2 | 1 | 6 | 3 | 2 | 5 | 1 | 2 | 3 | 3 | 4 | 3 | 1 | 3 | 44
  45-60 Years | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 2 | 1 | 2 | 1 | 1 | 0 | 3 | 4 | 2 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 12
  Male | 0 | 2 | 2 | 2 | 3 | 2 | 6 | 3 | 2 | 6 | 2 | 3 | 4 | 4 | 4 | 6 | 4 | 3 | 58
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 11
  Not Hispanic or Latino | 1 | 1 | 2 | 1 | 3 | 2 | 5 | 4 | 3 | 7 | 2 | 4 | 4 | 3 | 4 | 4 | 5 | 4 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) in PART-1: SAD
Description: An Adverse Event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were those with initial onset or increasing in severity between the first dose of study intervention and up to 36 days after last dose of study intervention. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. SAEs were adjudicated according to the investigator's assessment. Treatment-related AEs and SAEs were determined by the investigator.
Time Frame: Post the single dose of study intervention till up to 36 days
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Groups:
- Placebo (Suspension), Fasted: Participants received a single dose of placebo under fasted condition at 0 h
- Placebo (Suspension)/RTV 100 mg, Fasted: Participants received a single dose of placebo at 0 h under fasted condition in combination with RTV 100 mg at -12, 0 and 12h
- Placebo (Suspension)/RTV 100 mg, Fed: Participants received a single dose of placebo at 0 h under fed condition in combination with RTV 100 mg at -12, 0 and 12h
- PF-07321332 150 mg (Suspension), Fasted: Participants received a single dose of PF-07321332 150 mg (suspension) alone at 0 h under fasted condition
- PF-07321332 500 mg (Suspension), Fasted: Participants received a single dose of PF-07321332 500 mg (suspension) alone at 0 h under fasted condition
- PF-07321332 1500 mg (Suspension), Fasted: Participants received a single dose of PF-07321332 1500 mg (suspension) alone at 0 h under fasted condition
- PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted: Participants received a single dose of PF-07321332 250 mg (suspension) at 0 h under fasted condition in combination with RTV 100 mg at -12, 0 and 12h
- PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed: Participants received a single dose of PF-07321332 250 mg (suspension) at 0 h under fed condition in combination with RTV 100 mg at -12, 0 and 12h
- PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted: Participants received a single dose of PF-07321332 750 mg (suspension) at 0 h under fasted condition in combination with RTV 100 mg at -12, 0 and 12h
Arm/Group | Placebo (Suspension), Fasted | Placebo (Suspension)/RTV 100 mg, Fasted | Placebo (Suspension)/RTV 100 mg, Fed | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6 | 4 | 2 | 4 | 4 | 4 | 4 | 4 | 4
Participants
  Participants with all-causality TEAEs | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  Participants with treatment-related TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with all-causality SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with severe AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants discontinued from study due to AEs | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Discontinued study drug due to AE, study continued | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dose reduced/temporary discontinuation due to AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs in PART-1: SAD
Description: Vital signs (temperature, respiratory rate, pulse rate [PR], systolic blood pressure [SBP], and diastolic blood pressure [DBP]) were obtained with participants following at least 5 minutes of supine rest. Categorical criteria were defined as DBP: value <50 millimeters of mercury (mm Hg), increase >=20 mm Hg, or decrease >=20 mm Hg; PR: value <40 beats per minute (bpm) or value >120 bpm; SBP: value <90 mm Hg, increase >=30 mm Hg, or decrease >=30 mm Hg. Clinical significance of vital signs was determined at the investigator's discretion. The analysis population included all participants who received at least 1 dose of study intervention and had at least 1 assessment undertaken post treatment.
Time Frame: Baseline up to Day 2 of the final period
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Groups:
- Placebo (Suspension), Fasted: Participants received a single dose of placebo under fasted condition at 0 hour (h)
- Placebo (Suspension)/RTV 100 mg, Fasted: Participants received a single dose of placebo at 0 h under fasted condition in combination with ritonavir (RTV) 100 mg at -12, 0 and 12h
Arm/Group | Placebo (Suspension), Fasted | Placebo (Suspension)/RTV 100 mg, Fasted | Placebo (Suspension)/RTV 100 mg, Fed | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6 | 4 | 2 | 4 | 4 | 4 | 4 | 4 | 4
Participants
  SBP value <90 mmHg | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SBP decrease >=30 mmHg | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  DBP decrease >=20 mmHg | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Laboratory Abnormalities in PART-1: SAD
Description: Laboratory parameters included hematology, chemistry, urinalysis, and other (urine drug screening, Severe Acute Respiratory Syndrome Coronavirus 2 [SARS-CoV-2] reverse transcription polymerase chain reaction [RT-PCR], estimated glomerular filtration rate [eGFR], pregnancy test [beta human chorionic gonadotropin [b-hCG]], activated partial thromboplastin time [aPTT], prothrombin time [PT] - international normalized ratio [INR], fibrinogen, thyroid stimulating hormone [TSH], Free thyroxine [T4]). The clinical significance of laboratory parameters was determined at the investigator's discretion. The analysis population included all participants who received at least 1 dose of the study intervention.
Time Frame: Baseline up to Day 4 of the final period
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Arm/Group | Placebo (Suspension)/RTV 100 mg, Fasted | Placebo (Suspension)/RTV 100 mg, Fed | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 4 | 2 | 4 | 4 | 4 | 4 | 4 | 4
Participants | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 2

4. Primary Outcome: Number of Participants With TEAEs in PART-2:MAD
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were those with initial onset or increasing in severity between the first dose of study intervention and up to 36 days after last dose of study intervention. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. SAEs were adjudicated according to the investigator's assessment. Treatment-related AEs and SAEs were determined by the investigator.
Time Frame: Post first dose till up to 45 days after last dose of study intervention
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Groups:
- Placebo (Suspension)/RTV 100 mg BID, Fasted: Participants received placebo (suspension)/RTV 100 mg BID for 10 days under fasted condition
- PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted: Participants received PF-07321332/RTV 75/100 mg BID for 10 days under fasted condition
- PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted: Participants received PF-07321332 (suspension)/RTV 250/100 mg BID for 10 days under fasted condition
- PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted: Participants received PF-07321332 (suspension)/RTV 500/100 mg BID for 10 days under fasted condition
- Placebo (Suspension)/RTV 100 mg BID, Fasted, Japanese: Japanese participants received placebo (suspension)/RTV 100 mg BID for 10 days under fasted condition
- PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese: Japanese participants received PF-07321332 (suspension)/RTV 250/100 mg BID for 10 days under fasted condition
Arm/Group | Placebo (Suspension)/RTV 100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | Placebo (Suspension)/RTV 100 mg BID, Fasted, Japanese | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 8 | 4 | 4 | 7 | 2 | 4
Participants
  Participants with all-causality TEAEs | 4 | 3 | 3 | 4 | 2 | 4
  Participants with treatment-related TEAEs | 1 | 0 | 2 | 2 | 1 | 2
  Participants with all-causality SAEs | 0 | 0 | 0 | 0 | 0 | 0
  Participants with severe AEs | 0 | 0 | 0 | 0 | 0 | 0
  Participants discontinued from study due to AEs | 0 | 0 | 0 | 0 | 0 | 0
  Discontinued study drug due to AE, study continued | 0 | 0 | 0 | 0 | 0 | 0
  Dose reduced/temporary discontinuation due to AEs | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs in PART-2: MAD
Description: Vital signs (temperature, respiratory rate, PR, SBP, DBP) were obtained with participants following at least 5 minutes of supine rest. Categorical criteria were defined as DBP: value <50 mm Hg, increase >=20 mm Hg, or decrease >=20 mm Hg; PR: value <40 bpm or value >120 bpm; SBP: value <90 mm Hg, increase >=30 mm Hg, or decrease >=30 mm Hg. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Baseline up to Day 12
Population: The analysis population included all participants who received at least 1 dose of study intervention and had at least 1 assessment undertaken post treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Suspension)/RTV 100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | Placebo (Suspension)/RTV 100 mg BID, Fasted, Japanese | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 8 | 4 | 4 | 7 | 2 | 4
Participants
  SBP value <90 mmHg | 0 | 0 | 1 | 0 | 0 | 1
  SBP decrease >=30 mmHg | 0 | 0 | 0 | 0 | 1 | 0
  DBP value <50 mmHg | 1 | 0 | 0 | 0 | 0 | 1
  PR value <40 bpm | 0 | 0 | 0 | 1 | 0 | 0

6. Primary Outcome: Number of Participants With Laboratory Abnormalities in PART-2: MAD
Description: Laboratory parameters included hematology, chemistry, urinalysis, and other (urine drug screening, SARS-CoV-2 RT-PCR, eGFR, pregnancy test [b-hCG], aPTT, PT-INR, fibrinogen, TSH, Free T4). The clinical significance of laboratory parameters was determined at the investigator's discretion. The analysis population included all participants who received at least 1 dose of the study intervention.
Time Frame: Baseline up to Day 12
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Arm/Group | Placebo (Suspension)/RTV 100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | Placebo (Suspension)/RTV 100 mg BID, Fasted, Japanese | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 8 | 4 | 4 | 7 | 2 | 4
Participants | 5 | 2 | 4 | 5 | 2 | 3

7. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to The Time of The Last Quantifiable Concentration (AUClast) of Tablet Formulation and Suspension in PART-3: rBA/FE
Description: AUClast is area under the concentration-time profile from time 0 (pre-dose) to the time of the last quantifiable concentration.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: The analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- PF-07321332 250 mg (Suspension), Fasted: Participants received a single dose of PF-07321332 250 mg (suspension) under fasted condition
- PF-07321332 250 mg (Tablet), Fasted: Participants received a single dose of PF-07321332 250 mg (tablet) under fasted condition
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted
Number analyzed (Participants) | 12 | 12
nanogram*hour per milliliter (ng*hr/mL) | 3318 (35) | 2695 (46)
Statistical Analysis 1: Comparison: PF-07321332 250 mg (Suspension), Fasted vs PF-07321332 250 mg (Tablet), Fasted; Test type: Other — Natural log transformed AUClast for PF-07321332 was analyzed using a mixed effect model with sequence, period, and treatment included as fixed effects and subject nested within sequence as a random effect. PF-07321332 250 mg (Tablet), Fasted was the test treatment and PF-07321332 250 mg (Suspension), Fasted was the reference treatment; Ratio of Adjusted Geometric Means = 81.21, 90% CI 2-sided [69.21 to 95.28]

8. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of Tablet Formulation and Suspension in PART-3: rBA/FE
Description: AUCinf is area under the concentration-time profile from time 0 (pre-dose) extrapolated to infinite time. Natural log transformed AUCinf for PF-07321332 was analyzed to provide an estimate of the ratio of adjusted geometric means (Test [tablet] /Reference [suspension]) and 90% CI for the ratio.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/ml
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted
Number analyzed (Participants) | 7 | 9
ng*hr/ml | 3513 (38) | 2958 (50)
Statistical Analysis 1: Comparison: PF-07321332 250 mg (Suspension), Fasted vs PF-07321332 250 mg (Tablet), Fasted; Test type: Other — Natural log transformed AUCinf for PF-07321332 was analyzed using a mixed effect model with sequence, period, and treatment included as fixed effects and subject nested within sequence as a random effect. PF-07321332 250 mg (Tablet), Fasted was the test treatment and PF-07321332 250 mg (Suspension), Fasted was the reference treatment; Ratio of Adjusted Geometric Means = 76.06, 90% CI 2-sided [60.14 to 96.20]

9. Primary Outcome: Maximum Plasma Concentration (Cmax) of Tablet Formulation and Suspension in PART-3: rBA/FE
Description: Cmax is maximum plasma concentration. It was observed directly from data. Natural log transformed Cmax for PF-07321332 was analyzed to provide an estimate of the ratio of adjusted geometric means (Test [tablet] /Reference [suspension]) and 90% CI for the ratio.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted
Number analyzed (Participants) | 12 | 12
nanogram per milliliter (ng/mL) | 883.1 (37) | 497.8 (37)
Statistical Analysis 1: Comparison: PF-07321332 250 mg (Suspension), Fasted vs PF-07321332 250 mg (Tablet), Fasted; Test type: Other — Natural log transformed Cmax for PF-07321332 was analyzed using a mixed effect model with sequence, period, and treatment included as fixed effects and subject nested within sequence as a random effect. PF-07321332 250 mg (Tablet), Fasted was the test treatment and PF-07321332 250 mg (Suspension), Fasted was the reference treatment; Ratio of Adjusted Geometric Means = 56.38, 90% CI 2-sided [43.42 to 73.19]

10. Primary Outcome: Total Percent Recovery of Drug-Related Material in Urine in PART-4: ME
Description: Total recovery of drug-related material excreted in urine, expressed as a percent of total dose administered, measured by fluorine-19 nuclear magnetic resonance (19F-NMR).
Time Frame: Day 1 to Day 11
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: Percent of the dose
Groups:
- PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted: Participants received a single oral dose of PF-07321332 300 mg with RTV (4 doses of 100 mg at -12, 0, 12, and 24 hours relative to PF-07321332)
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
Percent of the dose
  PF-07321332-related material by 19F-NMR | 47.0 (10.3)
  M8 (PF-07331782) | 2.6 (1.1)

11. Primary Outcome: Total Percent Recovery of Drug-Related Material in Feces in PART-4: ME
Description: Total recovery of drug-related material excreted in feces, expressed as a percent of total dose administered, measured by 19F-NMR.
Time Frame: Day 1 to Day 11
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: Percent of the dose
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
Percent of the dose
  PF-07321332-related material by 19F-NMR | 33.7 (13.3)
  M8 (PF-07331782) | 1.6 (0.6)

12. Primary Outcome: Total Percent Recovery of Drug-Related Material in Excreta (Urine and Feces Combined) in PART-4: ME
Description: Total recovery of drug-related material excreted in urine and feces combined, expressed as a percent of total dose administered, measured by 19F-NMR.
Time Frame: Day 1 to Day 11
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: Percent of the dose
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
Percent of the dose
  PF-07321332-related material by 19F-NMR | 80.7 (8.0)
  M8 (PF-07331782) | 4.2 (1.3)
  Total | 84.9 (8.9)

13. Primary Outcome: Number of Participants With TEAEs in PART-5: SE
Description: as for outcome 4
Time Frame: Post first dose till up to 36 days after last dose of study intervention
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Groups:
- Placebo (Suspension)/RTV 100 mg: Participants received placebo with RTV (3 doses of 100 mg at -12, 0, and 12 hours relative to placebo)
- PF-07321332 2250 mg (Suspension)/RTV 100 mg: PF-07321332 2250 mg was administered as 3 split doses of 750 mg at 0, 2h and 4h, with RTV (3 doses of 100 mg at -12, 0 and 12 hours relative to PF-07321332).
Arm/Group | Placebo (Suspension)/RTV 100 mg | PF-07321332 2250 mg (Suspension)/RTV 100 mg
Number analyzed (Participants) | 10 | 10
Participants
  Participants with all-causality TEAEs | 3 | 3
  Participants with treatment-related TEAEs | 1 | 1
  Participants with all-causality SAEs | 0 | 0
  Participants with severe AEs | 0 | 0
  Participants discontinued from study due to AEs | 0 | 0
  Discontinued study drug due to AE, study continued | 0 | 0
  Dose reduced/temporary discontinuation due to AEs | 0 | 0

14. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs in PART-5: SE
Description: as for outcome 5
Time Frame: Baseline up to Day 5 of the final period
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Arm/Group | Placebo (Suspension)/RTV 100 mg | PF-07321332 2250 mg (Suspension)/RTV 100 mg
Number analyzed (Participants) | 10 | 10
Participants
  SBP value <90 mmHg | 1 | 0
  SBP decrease >= 30 mmHg | 1 | 1

15. Primary Outcome: Number of Participants With Laboratory Abnormalities in PART-5: SE
Description: as for outcome 6
Time Frame: Baseline up to Day 5 of the final period
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Arm/Group | Placebo (Suspension)/RTV 100 mg | PF-07321332 2250 mg (Suspension)/RTV 100 mg
Number analyzed (Participants) | 10 | 10
Participants | 1 | 2

16. Secondary Outcome: Cmax of Plasma PF-07321332 in PART-1: SAD
Description: Cmax is maximum plasma concentration. It was observed directly from data.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
ng/mL | 667.7 (28) | 674.4 (38) | 1538 (32) | 2882 (25) | 3323 (13) | 5086 (25)

17. Secondary Outcome: Time for Cmax (Tmax) of Plasma PF-07321332 in PART-1: SAD
Description: Time to reach Cmax.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hr
Arm/Group | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
hr | 0.634 [0.550 to 1.50] | 1.00 [0.517 to 1.00] | 1.00 [0.533 to 2.00] | 2.75 [1.50 to 4.00] | 4.00 [4.00 to 4.00] | 2.00 [1.50 to 4.00]

18. Secondary Outcome: AUClast of Plasma PF-07321332 in PART-1: SAD
Description: as for outcome 7
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
ng*hr/mL | 2125 (34) | 3753 (29) | 10870 (47) | 27600 (13) | 28020 (16) | 64230 (39)

19. Secondary Outcome: AUCinf of PF-07321332 in PART-1: SAD
Description: AUCinf is area under the concentration-time profile from time 0 (pre-dose) extrapolated to infinite time.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 3 | 2 | 0 | 4 | 4 | 4
ng*hr/mL | 2247 (42) | NA (NA) — Only individual values were reported: 5480 and 5450. |  | 28220 (14) | 28640 (17) | 66760 (45)

20. Secondary Outcome: Dose Normalized Cmax (Cmax[dn]) of Plasma PF-07321332 in PART-1: SAD
Description: Cmax is maximum plasma concentration. It was observed directly from data. Cmax(dn) = Cmax / dose.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
ng/mL/mg | 4.450 (28) | 1.349 (38) | 1.025 (32) | 11.53 (25) | 13.32 (13) | 6.782 (25)

21. Secondary Outcome: Dose Normalized AUCinf (AUCinf[dn]) of Plasma PF-07321332 in PART-1: SAD
Description: AUCinf is area under the concentration-time profile from time 0 (pre-dose) extrapolated to infinite time. AUCinf(dn) = AUCinf/dose.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 3 | 2 | 0 | 4 | 4 | 4
ng*hr/mL/mg | 14.97 (42) | NA (NA) — Only individual values were reported: 11 and 10.9. |  | 112.8 (14) | 114.2 (17) | 89.14 (45)

22. Secondary Outcome: Dose Normalized AUClast (AUClast[dn]) of Plasma PF-07321332 in PART-1: SAD
Description: AUClast is area under the concentration-time profile from time 0 (pre-dose) to the time of the last quantifiable concentration. AUClast(dn) = AUClast /dose.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
ng*hr/mL/mg | 14.15 (34) | 7.507 (29) | 7.247 (47) | 110.4 (13) | 112.0 (16) | 85.77 (40)

23. Secondary Outcome: Apparent Volume of Distribution (Vz/F) in PART-1: SAD
Description: Vz/F = Dose/(AUCinf*kel), where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 3 | 2 | 0 | 4 | 4 | 4
Liter | 190.6 (36) | NA (NA) — Only individual values were reported: 2440 and 3390. |  | 87.98 (28) | 73.48 (47) | 181.9 (35)

24. Secondary Outcome: Apparent Clearance (CL/F) in PART-1: SAD
Description: CL/F is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F = Dose/AUCinf.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour (L/hr)
Arm/Group | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 3 | 2 | 0 | 4 | 4 | 4
liter/hour (L/hr) | 66.83 (43) | NA (NA) — Only individual values were reported: 91.2 and 91.8. |  | 8.865 (14) | 8.735 (17) | 11.22 (45)

25. Secondary Outcome: Terminal Half-Life (t1/2) of Plasma PF-07321332 in PART-1: SAD
Description: t1/2 is the time measured for the plasma concentration of drug to decrease by one half of its initial concentration.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 3 | 2 | 0 | 4 | 4 | 4
hr | 2.023 (0.54556) | NA (NA) — Only individual values were reported: 18.5 and 25.6. |  | 6.935 (1.0794) | 6.005 (1.6502) | 12.86 (8.4196)

26. Secondary Outcome: Cmax of Plasma PF-07321332 in PART-2: MAD on Day 1, Day 5 and Day 10
Description: Cmax is maximum plasma concentration. It was observed directly from data.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose on Day 1, Day 5; and pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16 hours post-dose on Day 10.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
ng/mL
  Day 1 | 1042 (28) | 2435 (36) | 3051 (32) | 1925 (25)
  Day 5 | 2224 (27) | 4774 (21) | 5296 (21) | 3674 (28)
  Day 10 | 2055 (14) | 5123 (24) | 5607 (17) | 3772 (21)

27. Secondary Outcome: Tmax of Plasma PF-07321332 in PART-2: MAD on Day 1, Day 5 and Day 10
Description: Time to reach Cmax.
Time Frame: as for outcome 26
Population: as for outcome 7
Measure: Median (Full Range); unit: hr
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
hr
  Day 1 | 1.75 [1.00 to 2.00] | 1.50 [1.00 to 4.00] | 2.00 [1.50 to 2.17] | 2.75 [1.00 to 4.02]
  Day 5 | 1.00 [1.00 to 1.50] | 0.750 [0.500 to 1.50] | 1.50 [1.00 to 2.02] | 1.26 [1.00 to 2.02]
  Day 10 | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 2.00] | 1.50 [1.00 to 2.00] | 1.50 [0.500 to 2.02]

28. Secondary Outcome: Area Under the Plasma Concentration Time Profile From Time 0 to Time Tau (AUCtau) of Plasma PF-07321332 in PART-2: MAD on Day 1, Day 5 and Day 10
Description: AUCtau is area under the concentration-time profile from time 0 (pre-dose) to end of dosing interval, where dosing interval was 12 hours.
Time Frame: as for outcome 26
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
ng*hr/mL
  Day 1 | 6017 (33) | 18700 (43) | 22610 (37) | 13130 (26)
  Day 5 | 12570 (17) | 35560 (26) | 38150 (23) | 25480 (26)
  Day 10 | 12650 (16) | 37780 (27) | 39780 (20) | 26930 (15)

29. Secondary Outcome: Cmax(dn) of Plasma PF-07321332 in PART-2: MAD on Day 1, Day 5 and Day 10
Description: Cmax is maximum plasma concentration. It was observed directly from data. Cmax(dn) = Cmax / dose.
Time Frame: as for outcome 26
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
ng/mL/mg
  Day 1 | 13.89 (28) | 9.755 (36) | 6.103 (32) | 7.698 (25)
  Day 5 | 29.66 (27) | 19.10 (21) | 10.59 (21) | 14.70 (28)
  Day 10 | 27.40 (14) | 20.49 (25) | 11.22 (17) | 15.08 (21)

30. Secondary Outcome: Dose Normalized AUCtau (AUCtau[dn]) of Plasma PF-07321332 in PART-2: MAD on Day 1, Day 5 and Day 10
Description: AUCtau is area under the concentration-time profile from time 0 (pre-dose) to end of dosing interval, where dosing interval was 12 hours. AUCtau(dn) = AUCtau/dose.
Time Frame: as for outcome 26
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
ng*hr/mL/mg
  Day 1 | 80.19 (33) | 74.76 (43) | 45.23 (37) | 52.60 (26)
  Day 5 | 167.7 (17) | 141.9 (26) | 76.32 (23) | 102.0 (26)
  Day 10 | 168.3 (16) | 151.1 (26) | 79.56 (20) | 107.7 (15)

31. Secondary Outcome: Average Plasma Concentration Over the Dosing Interval (Cav) of Plasma PF-07321332 in PART-2: MAD on Day 5 and Day 10
Description: Cav is average plasma concentration over the dosing interval, where dosing interval was 12 hours.
Time Frame: as for outcome 26
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
ng/mL
  Day 5 | 1049 (17) | 2963 (26) | 3181 (23) | 2124 (26)
  Day 10 | 1053 (16) | 3147 (27) | 3314 (20) | 2245 (14)

32. Secondary Outcome: Minimum Observed Concentration During the Dosing Interval (Cmin) of Plasma PF-07321332 in PART-2: MAD on Day 5 and Day 10
Description: Cmin is minimum observed concentration during the dosing interval, where dosing interval was 12 hours.
Time Frame: as for outcome 26
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
ng/mL
  Day 5 | 251.0 (11) | 1315 (37) | 1195 (29) | 707.3 (35)
  Day 10 | 245.3 (27) | 1480 (27) | 1279 (31) | 12.50 (NA) — Zero values had been substituted with 0.0001 prior to log transformation

33. Secondary Outcome: Observed Accumulation Ratio for AUCtau (Rac) Plasma PF-07321332 in PART-2: MAD on Day 5 and Day 10
Description: Rac was calculated as Day 5 or Day 10 AUCtau/Day 1 AUCtau.
Time Frame: as for outcome 26
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
Ratio
  Day 5 | 2.091 (24) | 1.901 (22) | 1.685 (29) | 1.937 (18)
  Day 10 | 2.104 (30) | 2.022 (16) | 1.757 (26) | 2.047 (16)

34. Secondary Outcome: Observed Accumulation Ratio for Cmax (Rac,Cmax) of Plasma PF-07321332 in PART-2: MAD on Day 5 and Day 10
Description: Rac,Cmax is Day 5 or Day 10 Cmax/Day 1 Cmax.
Time Frame: as for outcome 26
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
Ratio
  Day 5 | 2.133 (25) | 1.959 (16) | 1.733 (24) | 1.909 (26)
  Day 10 | 1.971 (34) | 2.101 (16) | 1.840 (29) | 1.962 (14)

35. Secondary Outcome: Peak-to-Trough Ratio (PTR) of Plasma PF-07321332 in PART-2: MAD on Day 5 and Day 10
Description: PTR is defined as peak-to-trough ratio. PTR = Cmax/Cmin.
Time Frame: as for outcome 26
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
Ratio
  Day 5 | 8.857 (27) | 3.635 (21) | 4.430 (14) | 5.194 (19)
  Day 10 | 8.383 (16) | 3.462 (5) | 4.385 (17) | 6.270 (32)

36. Secondary Outcome: CL/F of Plasma PF-07321332 in PART-2:MAD on Day 5 and Day 10
Description: CL/F is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F = Dose/AUCtau.
Time Frame: as for outcome 26
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
L/hr
  Day 5 | 5.966 (17) | 7.032 (26) | 13.11 (23) | 9.814 (26)
  Day 10 | 5.933 (16) | 6.617 (27) | 12.57 (20) | 9.278 (15)

37. Secondary Outcome: Vz/F of Plasma PF-07321332 in PART-2: MAD on Day 10
Description: Vz/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F = Dose/(AUCinf*kel), where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16 hours post-dose on Day 10.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
Liter | 66.43 (24) | 63.40 (13) | 142.4 (37) | 65.04 (31)

38. Secondary Outcome: t1/2 of of Plasma PF-07321332 in PART-2: MAD on Day 10
Description: t1/2 is the time measured for the plasma concentration of drug to decrease by one-half of its initial concentration.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16 hours post-dose on Day 10.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
hr | 7.955 (2.0401) | 6.795 (1.7072) | 8.047 (1.7871) | 5.163 (2.0915)

39. Secondary Outcome: Amount Excreted in Urine as Unchanged Drug Over the Dosing Interval Tau (Aetau) in PART-2: MAD on Day 10
Description: Ae is the cumulative amount of drug recovered unchanged in urine during the dosing interval, where the dosing interval is 12 hours. Aetau is the sum of (urine volume × urine concentration) for each collection over the dosing interval.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16 hours post-dose on Day 10.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
mg | 47.83 (12) | 129.9 (4) | 116.5 (122) | 135.4 (5)

40. Secondary Outcome: Percent of Dose Excreted in Urine as Unchanged Drug Over the Dosing Interval Tau (Aetau%) in PART-2: MAD on Day 10
Description: Aetau% is defined as percent of dose excreted in urine as unchanged drug over the dosing interval, where the dosing interval is 12 hours. Aetau% = Aetau / Dose * 100.
Time Frame: Pre-dose to 12 hours post-dose on Day 10
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
percentage of dose | 63.79 (12) | 51.81 (4) | 23.35 (121) | 54.20 (5)

41. Secondary Outcome: Renal Clearance (CLr) in PART-2: MAD on Day 10
Description: CLr is defined as the renal clearance. CLr = Aetau / AUCtau, where the dosing interval was 12 hours.
Time Frame: Pre-dose to 12 hours post-dose on Day 10
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese
Number analyzed (Participants) | 4 | 4 | 7 | 4
L/hr | 3.782 (20) | 3.433 (23) | 2.934 (128) | 5.028 (11)

42. Secondary Outcome: AUClast of Plasma PF-07321332 of Tablet Formulation Under Fed Condition and Fasted Condition in PART-3: rBA/FE
Description: AUClast is area under the concentration-time profile from time 0 (pre-dose) to the time of the last quantifiable concentration. Natural log transformed AUClast for PF-07321332 was analyzed to provide an estimate of the ratio of adjusted geometric means (Test [tablet under fed condition] /Reference [tablet under fasted condition]) and 90% CI for the ratio.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- PF-07321332 250 mg (Tablet), Fed: Participants received a single dose of PF-07321332 250 mg (tablet) under fed condition
Arm/Group | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 2695 (46) | 4012 (27)
Statistical Analysis 1: Comparison: PF-07321332 250 mg (Tablet), Fasted vs PF-07321332 250 mg (Tablet), Fed; Test type: Other — Natural log transformed AUClast for PF-07321332 was analyzed using a mixed effect model with sequence, period, and treatment included as fixed effects and subject nested within sequence as a random effect. PF-07321332 250 mg (Tablet), Fed was the test treatment and PF-07321332 250 mg (Tablet), Fasted was the reference treatment; Ratio of Adjusted Geometric Means = 148.91, 90% CI 2-sided [126.92 to 174.72]

43. Secondary Outcome: AUCinf of Plasma PF-07321332 of Tablet Formulation Under Fed Condition and Fasted Condition in PART-3: rBA/FE
Description: AUCinf is area under the concentration-time profile from time 0 (pre-dose) extrapolated to infinite time. Natural log transformed AUCinf for PF-07321332 was analyzed to provide an estimate of the ratio of adjusted geometric means (Test [tablet under fed condition] /Reference [tablet under fasted condition]) and 90% CI for the ratio.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed
Number analyzed (Participants) | 9 | 9
ng*hr/mL | 2958 (50) | 4256 (24)
Statistical Analysis 1: Comparison: PF-07321332 250 mg (Tablet), Fasted vs PF-07321332 250 mg (Tablet), Fed; Test type: Other — Natural log transformed AUCinf for PF-07321332 was analyzed using a mixed effect model with sequence, period, and treatment included as fixed effects and subject nested within sequence as a random effect. PF-07321332 250 mg (Tablet), Fed was the test treatment and PF-07321332 250 mg (Tablet), Fasted was the reference treatment; Ratio of Adjusted Geometric Means = 146.80, 90% CI 2-sided [118.80 to 181.41]

44. Secondary Outcome: Cmax of Plasma PF-07321332 of Tablet Formulation Under Fed Condition and Fasted Condition in PART-3: rBA/FE
Description: Cmax is maximum plasma concentration. It was observed directly from data. Natural log transformed Cmax for PF-07321332 was analyzed to provide an estimate of the ratio of adjusted geometric means (Test [tablet under fed condition] /Reference [tablet under fasted condition]) and 90% CI for the ratio.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12
ng/mL | 497.8 (37) | 1219 (55)
Statistical Analysis 1: Comparison: PF-07321332 250 mg (Tablet), Fasted vs PF-07321332 250 mg (Tablet), Fed; Test type: Other — Natural log transformed Cmax for PF-07321332 was analyzed using a mixed effect model with sequence, period, and treatment included as fixed effects and subject nested within sequence as a random effect. PF-07321332 250 mg (Tablet), Fed was the test treatment and PF-07321332 250 mg (Tablet), Fasted was the reference treatment; Ratio of Adjusted Geometric Means = 244.84, 90% CI 2-sided [188.58 to 317.87]

45. Secondary Outcome: Cmax(dn) of Plasma PF-07321332 in PART-3: rBA/FE
Description: Cmax is maximum plasma concentration. It was observed directly from data. Cmax(dn) = Cmax / dose.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 12
ng/mL/mg | 3.533 (37) | 1.992 (37) | 4.874 (55)

46. Secondary Outcome: Tmax of Plasma PF-07321332 in PART-3: rBA/FE
Description: Time to reach Cmax.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hr
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 12
hr | 1.00 [0.500 to 4.00] | 1.00 [0.500 to 4.00] | 1.75 [0.500 to 4.00]

47. Secondary Outcome: AUClast(dn) of Plasma PF-07321332 in PART-3: rBA/FE
Description: as for outcome 22
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 12
ng*hr/mL/mg | 13.27 (35) | 10.78 (46) | 16.03 (27)

48. Secondary Outcome: AUCinf(dn) of Plasma PF-07321332 in PART-3: rBA/FE
Description: as for outcome 21
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed
Number analyzed (Participants) | 7 | 9 | 9
ng*hr/mL/mg | 14.06 (38) | 11.82 (50) | 17.03 (24)

49. Secondary Outcome: CL/F of Plasma PF-07321332 in PART-3: rBA/FE
Description: CL/F is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F = Dose/AUCinf.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed
Number analyzed (Participants) | 7 | 9 | 9
L/hr | 71.07 (38) | 84.56 (50) | 58.70 (24)

50. Secondary Outcome: Vz/F of Plasma PF-07321332 in PART-3: rBA/FE
Description: as for outcome 23
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed
Number analyzed (Participants) | 7 | 9 | 9
Liter | 493.7 (63) | 1004 (41) | 151.0 (36)

51. Secondary Outcome: t1/2 of Plasma PF-07321332 in PART-3: rBA/FE
Description: t1/2 is the time measured for the plasma concentration of drug to decrease by one-half of its initial concentration.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, and 48 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed
Number analyzed (Participants) | 7 | 9 | 9
hr | 5.626 (3.0407) | 9.086 (4.1570) | 1.854 (0.55166)

52. Secondary Outcome: Number of Participants With TEAEs in PART-3: rBA/FE
Description: as for outcome 4
Time Frame: Post the single dose of study intervention till up to 36 days
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Participants with all-causality TEAEs | 3 | 3 | 1
  Participants with treatment-related TEAEs | 2 | 1 | 0
  Participants with all-causality SAEs | 0 | 0 | 0
  Participants with severe AEs | 0 | 0 | 0
  Participants discontinued from study due to AEs | 0 | 0 | 0
  Discontinued study drug due to AE, study continued | 0 | 0 | 0
  Dose reduced/temporary discontinuation due to AEs | 0 | 0 | 0

53. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities in PART-3: rBA/FE
Description: as for outcome 6
Time Frame: Baseline up to Day 3
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Arm/Group | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fed | PF-07321332 250 mg (Tablet), Fasted
Number analyzed (Participants) | 4 | 4 | 4
Participants | 1 | 2 | 0

54. Secondary Outcome: Cmax of Plasma PF-07321332 in PART-4: ME
Description: Cmax is maximum plasma concentration. It was observed directly from data.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
ng/mL | 4068 (14)

55. Secondary Outcome: Tmax of Plasma PF-07321332 in PART-4: ME
Description: Tmax is time to reach Cmax.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hr
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
hr | 2.00 [1.00 to 2.00]

56. Secondary Outcome: AUClast of Plasma PF-07321332 in PART-4: ME
Description: as for outcome 7
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
ng*hr/mL | 32960 (23)

57. Secondary Outcome: AUCinf of Plasma PF-07321332 in PART-4: ME
Description: AUCinf is area under the concentration-time profile from time 0 (pre-dose) extrapolated to infinite time.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
ng*hr/mL | 33470 (22)

58. Secondary Outcome: CL/F of Plasma PF-07321332 in PART-4: ME
Description: CL/F is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F = Dose/AUCinf.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
L/hr | 8.968 (22)

59. Secondary Outcome: Vz/F of Plasma PF-07321332 in PART-4: ME
Description: as for outcome 23
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
Liter | 115.8 (48)

60. Secondary Outcome: t1/2 of Plasma PF-07321332 in PART-4: ME
Description: t1/2 is the time measured for the plasma concentration of drug to decrease by one-half of its initial concentration.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
hr | 9.485 (3.1833)

61. Secondary Outcome: Number of Participants With TEAEs in PART-4: ME
Description: as for outcome 4
Time Frame: Post the single dose of study intervention till up to 36 days
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
Participants
  Participants with all-causality TEAEs | 1
  Participants with treatment-related TEAEs | 0
  Participants with all-causality SAEs | 0
  Participants with severe AEs | 0
  Participants discontinued from study due to AEs | 0
  Discontinued study drug due to AE, study continued | 0
  Dose reduced/temporary discontinuation due to AEs | 0

62. Secondary Outcome: Number of Participants With Laboratory Abnormalities in PART-4: ME
Description: Laboratory parameters included hematology, chemistry, urinalysis, and other (urine drug screening, SARS-CoV-2 RT-PCR, eGFR, pregnancy test [b-hCG], aPTT, PT-INR, fibrinogen, TSH, Free T4). The clinical significance of laboratory parameters was determined at the investigator's discretion.
Time Frame: Baseline up to Day 11
Population: The analysis population included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Arm/Group | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted
Number analyzed (Participants) | 6
Participants | 3

63. Secondary Outcome: Cmax of Plasma PF-07321332 in PART-5: SE
Description: Cmax is maximum plasma concentration. It was observed directly from data.
Time Frame: Pre-dose, 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-07321332 2250 mg (Suspension)/RTV 100 mg
Number analyzed (Participants) | 10
ng/mL | 15940 (27)

64. Secondary Outcome: Tmax of Plasma PF-07321332 in PART-5: SE
Description: Time to reach Cmax.
Time Frame: Pre-dose, 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hr
Arm/Group | PF-07321332 2250 mg (Suspension)/RTV 100 mg
Number analyzed (Participants) | 10
hr | 5.00 [3.02 to 6.03]

65. Secondary Outcome: AUClast of Plasma PF-07321332 in PART-5: SE
Description: as for outcome 7
Time Frame: Pre-dose, 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/ml
Arm/Group | PF-07321332 2250 mg (Suspension)/RTV 100 mg
Number analyzed (Participants) | 10
ng*hr/ml | 188200 (35)

66. Secondary Outcome: AUCinf of Plasma PF-07321332 in PART-5: SE
Description: AUCinf is area under the concentration-time profile from time 0 (pre-dose) extrapolated to infinite time.
Time Frame: Pre-dose, 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/ml
Arm/Group | PF-07321332 2250 mg (Suspension)/RTV 100 mg
Number analyzed (Participants) | 10
ng*hr/ml | 188800 (35)

67. Secondary Outcome: t1/2 of Plasma PF-07321332 in PART-5: SE
Description: t1/2 is the time measured for the plasma concentration of drug to decrease by one-half of its initial concentration.
Time Frame: Pre-dose, 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-07321332 2250 mg (Suspension)/RTV 100 mg
Number analyzed (Participants) | 10
hr | 7.450 (2.9357)

ADVERSE EVENTS:
Time Frame: Post first dose till up to 45 days after the last dose of the study intervention, up to 57 days.
Arm/Group | Placebo (Suspension), Fasted | Placebo (Suspension)/RTV 100 mg, Fasted | Placebo (Suspension)/RTV 100 mg, Fed | PF-07321332 150 mg (Suspension), Fasted | PF-07321332 500 mg (Suspension), Fasted | PF-07321332 1500 mg (Suspension), Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted | Placebo (Suspension)/RTV 100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted | Placebo (Suspension)/RTV 100 mg BID, Fasted, Japanese | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese | PF-07321332 250 mg (Suspension), Fasted | PF-07321332 250 mg (Tablet), Fasted | PF-07321332 250 mg (Tablet), Fed | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted | Placebo (Suspension)/RTV 100 mg | PF-07321332 2250 mg (Suspension)/RTV 100 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/2 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/8 | 0/4 | 0/4 | 0/7 | 0/2 | 0/4 | 0/12 | 0/12 | 0/12 | 0/6 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/2 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/8 | 0/4 | 0/4 | 0/7 | 0/2 | 0/4 | 0/12 | 0/12 | 0/12 | 0/6 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/6 | 1/4 | 1/2 | 0/4 | 1/4 | 1/4 | 1/4 | 0/4 | 0/4 | 4/8 | 3/4 | 3/4 | 4/7 | 2/2 | 4/4 | 3/12 | 3/12 | 1/12 | 1/6 | 3/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Suspension), Fasted (N=6) | Placebo (Suspension)/RTV 100 mg, Fasted (N=4) | Placebo (Suspension)/RTV 100 mg, Fed (N=2) | PF-07321332 150 mg (Suspension), Fasted (N=4) | PF-07321332 500 mg (Suspension), Fasted (N=4) | PF-07321332 1500 mg (Suspension), Fasted (N=4) | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fasted (N=4) | PF-07321332 250 mg (Suspension)/RTV 100 mg, Fed (N=4) | PF-07321332 750 mg (Suspension)/RTV 100 mg, Fasted (N=4) | Placebo (Suspension)/RTV 100 mg BID, Fasted (N=8) | PF-07321332 (Suspension)/RTV 75/100 mg BID, Fasted (N=4) | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted (N=4) | PF-07321332 (Suspension)/RTV 500/100 mg BID, Fasted (N=7) | Placebo (Suspension)/RTV 100 mg BID, Fasted, Japanese (N=2) | PF-07321332 (Suspension)/RTV 250/100 mg BID, Fasted, Japanese (N=4) | PF-07321332 250 mg (Suspension), Fasted (N=12) | PF-07321332 250 mg (Tablet), Fasted (N=12) | PF-07321332 250 mg (Tablet), Fed (N=12) | PF-07321332 300 mg (Suspension)/RTV 100 mg, Fasted (N=6) | Placebo (Suspension)/RTV 100 mg (N=10) | PF-07321332 2250 mg (Suspension)/RTV 100 mg (N=10)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT04756531/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT04756531/SAP_001.pdf